CLINICAL TRIAL: NCT01556295
Title: Assessment of Gesture Behavior and Knowledge on Low Back Pain Among Nurses
Brief Title: Gesture Behavior and Knowledge on Low Back Pain Among Nurses
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Federal University of São Paulo (Other)
Responsible Party: Principal Investigator, Hisa Costa Morimoto, Principal investigator, Federal University of São Paulo
Other Study IDs: 1586/08
Record Dates: First submitted 2012-03-13; First posted 2012-03-16 (Estimated); Last update posted 2012-03-19 (Estimated); Status verified 2012-03

CONDITIONS: Low Back Pain
Keywords: Nurses; Low back pain; Gesture behavior; Knowlegde
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Experimental
- Control

SUMMARY:
The aim of the proposed study is to evaluate knowledge on low back pain and gesture behavior among nurses with low back pain using validated measures and compare the findings to those from nurses without back pain.

DETAILED DESCRIPTION:
A controlled, cross-sectional study will be carried out with 100 nurses (50 with low back pain and 50 without low back pain). The following assessment measures will be employed: Visual analogue scale (VAS) for pain, Gesture Behavior Test (GBT), Low Back Pain Knowledge Questionnaire (LKQ), Roland Morris Questionnaire and the SF-36.

ELIGIBILITY:
Inclusion Criteria:

* Non-specific chronic low back pain,
* Performance in the hospital sector (hospitals, emergency rooms and/or intensive care units,
* Hourly load of at least 6 hours per day,
* Low back pain on most days in the last three months,
* Pain greater than 3 cm in visual analog scale (VAS).

Exclusion Criteria:

* Dispute,
* Previous surgery of the spine,
* Pregnant.

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Nurses with non-specific low back pain and healthy nurses
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2012-03; Primary Completion 2012-08 (Estimated); Study Completion 2013-04 (Estimated)

PRIMARY OUTCOMES:
Gesture behavior | One week

SECONDARY OUTCOMES:
Knowledge among low back pain | One week
Roland Morris Questionnaire | One week
  Used health status measure for low back pain
SF-36 | One week
  Quality of life by SF-36
Visual analogue scale (VAS) for pain | One week
  Evaluation pain

CONTACTS AND LOCATIONS:
Overall Officials: Hisa Morimoto, PT, Principal Investigator — Federal University of São Paulo; Anamaria Jones, PT, PHD, Study Director — Federal University of São Paulo; Jamil Natour, MD, PHD, Study Chair — Division of Rheumatology, Federal University of Sao Paulo
Locations (1):
- HIsa Costa Morimoto, São Paulo, São Paulo, Brazil

REFERENCES:
- [Background] Furtado R, Jones A, Furtado RN, Jennings F, Natour J. Validation of the Brazilian-Portuguese version of the Gesture Behavior Test for patients with non-specific chronic low back pain. Clinics (Sao Paulo). 2009;64(2):83-90. doi: 10.1590/s1807-59322009000200004. PMID 19219312
- [Derived] Morimoto HC, Jones A, Natour J. Assessment of gesture behavior and knowledge on low back pain among nurses. Adv Rheumatol. 2018 Sep 7;58(1):27. doi: 10.1186/s42358-018-0029-5. PMID 30657083
- See also: low back pain with rehabilitation — http://www.projetodiretrizes.org.br/projeto_diretrizes/072.pdf